CLINICAL TRIAL: NCT05085665
Title: Loiasis Cross-reactive Antigenemia and Treatment-related Adverse Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Center for Research on Filariasis and Other Tropical Diseases, Cameroon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201909003(2)
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Loiasis
MeSH Terms: conditions — Loiasis | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ivermectin (Experimental): All eligible participants received a single dose (150 ug/kg) ivermectin by mouth
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — single dose, 150 ug/kg

SUMMARY:
This study seeks to determine which Loa loa antigens are released into circulation when infected individuals are treated with ivermectin.

DETAILED DESCRIPTION:
A cohort of up to 50 participants with Loa loa microfilarial levels between 5,000 and 18,000 per ml/blood will be treated with ivermectin in an inpatient setting. Participants will be monitored for treatment-related adverse events for seven days post-treatment, and will have blood drawn on days 0, 1, 2, 3, and 7 post-treatment to assess for microfilarial load, cytokine, and antigen levels.

ELIGIBILITY:
Inclusion Criteria:

* Loa loa blood microfilariae of between 5,000 - 18,000 per mL

Exclusion Criteria:

* known allergy to ivermectin; severe comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur les Filarioses et autres Maladies Tropicales (CRFilMT), Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: potential participants were identified via screening for daytime L. loa Mf counts in communities in the Awae Health District
Pre-assignment Details: 41 participants were enrolled; 2 were excluded at the initial study visit: one for L. loa Mf counts >20,000 / mL blood and one due to concerns for significant past medical history
Period: Overall Study
Arm/Group | Ivermectin
Started | 41
Completed | 39
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ivermectin
Number analyzed (Participants) | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [44 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Cameroon | 39

OUTCOME MEASURES:

1. Primary Outcome: Cross-reactive Antigenemia
Description: N of participants with detectable Loa loa antigens in sera that cross-react with diagnostic tests for lymphatic filariasis (Filariasis Test Strip) on either day 1, 2, 3, or 7 post-treatment
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin
Number analyzed (Participants) | 39
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse events were assessed on days 1 - 7 post-treatment
Arm/Group | Ivermectin
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 34/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin (N=39)
asthenia (General disorders) | 13 (13) — asthenia (French): weakness / fatigue
fever (General disorders) | 7 (7)
itching (Skin and subcutaneous tissue disorders) | 11 (11) — pruritus, prurit(French)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
blurry vision (Eye disorders) | 4 (4) — vision floue (French)
decreased appetite (Gastrointestinal disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 8 (8)
vomiting (Gastrointestinal disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
abdominal pain (Gastrointestinal disorders) | 5 (5)
headache (General disorders) | 11 (11)
myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
lightheadedness (General disorders) | 5 (5)
cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
adenopathy (Immune system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT05085665/Prot_SAP_ICF_000.pdf